CLINICAL TRIAL: NCT00546026
Title: Does Mid-Gestation Placental Function Assessment Reduce Psychological Distress in Women With High-Risk Pregnancies?
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Ontario Mental Health Foundation (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sloan01
Record Dates: First submitted 2007-10-16; First posted 2007-10-18 (Estimated); Last update posted 2007-10-18 (Estimated); Status verified 2007-10

CONDITIONS: High-Risk Pregnancy
Keywords: placental function; high-risk pregnancies; psychological distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active group (Active Comparator): Receive assessment of placental function
  Interventions: Other: placental function assessment

INTERVENTIONS:
Other: placental function assessment — Formal assessment of placental function in mid-gestation by placental morphology and uterine artery Doppler at 20-22 weeks and re-interpretation of prior biochemical tests for Down's syndrome and spina bifida.

SUMMARY:
Women whose pregnancies are at judged to be at risk of a poor outcome from an early delivery due to medical problems such as diabetes or high blood pressure, are often very anxious during pregnancy, at least until they know they have passed the risk period of premature birth (after 8 months). Anxiety itself can have a significant effect on the developing baby, on the newborn child and the mother-infant bonding process. We will use a combination of pregnancy blood tests and an ultrasound assessment to check on placental function, since placental damage is the greatest cause of poor outcome. Most women tested this way will have normal results, and so may feel reassured and do better in pregnancy than untested women. The benefits may extend after birth to mother-infant bonding, breastfeeding success and a reduced risk of postnatal depression. We will randomly select an equal number of women for testing and no testing (like tossing a coin, known as a randomized control trial) to be confident that any benefits observed are genuine. The potential benefits of our research would be substantial for the mental health of many pregnant women, for their newborn and for their children as they grow up. The tests are easy to do and would add very little in terms of a woman's and in terms of the total costs of prenatal care.

DETAILED DESCRIPTION:
Women whose pregnancies are considered "high-risk" for medical reasons such (e.g. preeclampsia, coagulation problems), often develop anxiety because of the possibility of a poor outcome. Such anxiety can affect fetal development, neonatal wellbeing, child development and maternal mental health but it often goes unrecognized. Also, women are often reluctant to use medications during pregnancy, especially if they perceive there may be the slightest risk to the fetus. By assessing placental function at mid-pregnancy in this population, we can provide an accurate estimate of which women will develop severe complications later in the pregnancy. We propose to perform a pilot randomized control trial formally incorporating placental assessment (Doppler ultrasound of the uterine artery and reassessment of diagnostic tests done earlier in pregnancy), with one group of "high-risk" women receiving the intervention (followed by feedback). Measures of pregnancy outcome and anxiety will be compared with a control group receiving standard "high-risk" pregnancy care. Levels of anxiety will be measured throughout the pregnancy using standardized scales. We hypothesize that placental function testing will reduce the burden of anxiety for the majority of women who test negative in the placental assessment arm and that these women will have improved outcomes and measures of anxiety during and following pregnancy in comparison with untested women who perceive themselves to be at risk of pregnancy complications throughout pregnancy. We also anticipate that the outcome of the pregnancy in women in the "tested" group will be more favorable (e.g. reduced admissions of neonate to NICU).

ELIGIBILITY:
Inclusion Criteria:

* Patient of maternal/fetal medicine unit Mount Sinai Hospital
* Over 18 years of age
* Able to understand the nature of the study
* Able to provide consent to participation
* Singleton pregnancy
* Normal karyotype
* No major anatomical malformations at the 19 week ultrasound
* Fluent in English

Exclusion Criteria:

* Currently suffering from a major psychiatric illness or current use of psychotropic medications
* Current illegal substance or alcohol abuse
* Presence of a significant fetal structural abnormality on the 19 week ultrasound
* Abnormal karyotype
* Multifetal pregnancy

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure is STAI - The State Trait Anxiety Inventory | Cross-sectional

SECONDARY OUTCOMES:
Women who undergo the placental function assessment will deliver at a later gestation age, have less complications and stillbirths than untested women. Neonates will have higher APGAR scores at 1 and 5 minutes and less likely to be admitted to the NICU. | Cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Eileen P. Sloan, MD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada